CLINICAL TRIAL: NCT02712177
Title: Interaction Between Meningococcal Serogroup B Vaccine (Bexsero™) and Routine Infant Vaccines on the Risk of Occurrence and Recurrence of Adverse Events Following Immunization.
Brief Title: Bexsero™and Routine Infant Vaccines: Effect of Coadministration on the Safety of Immunization
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: GlaxoSmithKline (Industry); Canadian Immunization Research Network (Network)
Responsible Party: Principal Investigator, Gaston De Serres, Researcher, MD, PhD, CHU de Quebec-Universite Laval
Other Study IDs: 1224; 1224 (Other: Clinical Study Data request)
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Meningococcal Infections
Keywords: vaccine safety; interaction
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Heptavalent Pneumococcal Conjugate Vaccine; Priorix-Tetra vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Coadministration B_RV246: Subjects in this group received 4CMenB vaccine at 2, 4, and 6 months of age, administered concomitantly with routine infant vaccinations (Infanrix Hexa+Prevenar).
  Interventions: Biological: 4CMenb; Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB; Biological: conjugated pneumococcal vaccine
- Coadministration B_RV234: Subjects in this group received 4CMenB vaccine at 2, 3 and 4 months of age, administered concomitantly with routine infant vaccinations (Infanrix Hexa+Prevenar)..
  Interventions: Biological: 4CMenb; Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB; Biological: conjugated pneumococcal vaccine
- Coadministration B_MMRV12: Subjects in this group previously received three doses of 4CMenB and routine vaccine at 2, 4 and 6 months of age,respectively. They also received a booster (fourth) dose at 12 months of age concomitantly with one dose of MMRV vaccine.
  Interventions: Biological: 4CMenb; Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB; Biological: conjugated pneumococcal vaccine; Biological: MMRV
- Separate administration B246_RV357: Subjects in this group received 4CMenB vaccine at 2, 4, and 6 months of age; routine infant vaccinations (Infanrix Hexa+Prevenar) were administered at 3, 5 and 7 months of age.
  Interventions: Biological: 4CMenb; Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB; Biological: conjugated pneumococcal vaccine
- Separate administration B12_MMRV13: Subjects in this group previously received three doses of 4CMenB and routine vaccines (Infanrix Hexa+Prevenar) at 2, 4 and 6 months of age. They also received a booster (fourth) dose of 4CMenB at 12 months of age and one dose of MMRV vaccine at 13 months of age.
  Interventions: Biological: 4CMenb; Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB; Biological: conjugated pneumococcal vaccine; Biological: MMRV
- Routine vaccines only at 2, 3 and 4 months of age (RV234): Subjects in this group received routine infant vaccines (Infanrix Hexa+Prevenar) at 2, 3 and 4 months of age.
  Interventions: Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB; Biological: conjugated pneumococcal vaccine
- Routine vaccines only at 2, 4 and 6 months of age.(RV246): Subjects in this group received routine infant vaccines (Infanrix Hexa+Prevenar) at 2, 4 and 6 months of age.
  Interventions: Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB; Biological: conjugated pneumococcal vaccine

INTERVENTIONS:
Biological: 4CMenb
  Other Names: Bexsero
  Groups: Coadministration B_MMRV12; Coadministration B_RV234; Coadministration B_RV246; Separate administration B12_MMRV13; Separate administration B246_RV357
Biological: diphtheria,tetanus,pertussis+polio+Hepatitis B+HiB
  Other Names: Infanrix Hexa
Biological: conjugated pneumococcal vaccine
  Other Names: Prevenar
Biological: MMRV
  Other Names: Priorix Tetra
  Groups: Coadministration B_MMRV12; Separate administration B12_MMRV13

SUMMARY:
Bexsero™ is a four component serogroup B meningococcal vaccine (4CMenB) licensed in Europe, Canada, and Australia in 2014. Prelicensure studies and post marketing surveillance data showed that 4CMenB has a high reactogenicity especially when coadministered with other infant routine vaccines [1-2]. While this suggests that coadministration causes an interaction resulting in a greater risk of adverse events following Immunization (AEFI) only the AEFI after the 4CMenB dose and not those occurring after routine vaccine immunizations were reported, underestimating the total risk associated with immunization at separate visits. For financial and practical reasons, coadministration of infant vaccines is preferred to separate visits. Separate visits may however be preferred if the sum of the AEFI risk at each visit is significantly smaller than the risk with coadministration and/or if the AEFI has a lesser severity. The purpose of this study is to recalculate the risk of occurrence and severity of AEFI with the coadministration of Bexsero™ and routine vaccines compared to separate injections to assess the interaction occurring with co-administration. Investigators will also estimate the risk of recurrence of AEFI at subsequent immunizations with the 4CMenB and assess if this risk varies with separate or coadministration with routine vaccines. To achieve these purposes, investigators will perform a secondary analysis of the data of three randomized controlled trials (clinicaltrials.gov identifiers: NCT00657709, NCT00847145 and NCT00721396) that evaluated 5025 children aged 2 to 14 months of whom 4535 were randomized to receive 3 to 4 doses of 4CMenB concomitantly or alternatively with routine vaccinations (DTaP-Inactivated polio virus -HepatitisB/Haemophilus influenzae type b [Infanrix Hexa™], Pneumococcal conjugate vaccine, 7 valent [Prevenar™] or Measles-Mumps-Rubella-Varicella vaccine [Priorix-Tetra™]) [1,2].

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month old infants (55-89 days, inclusive), who were born after full term pregnancy with an estimated gestational age ≥ 37 weeks
* Parent/legal guardian has given written informed consent after the nature of the study has been explained.

Main exclusion Criteria :

* History of any meningococcal B or C vaccine administration; prior vaccination with routine infant vaccines (Diphtheria, Tetanus, Pertussis, Polio, Haemophilus influenzae type b (Hib), and Pneumococcal antigens);
* Previous ascertained or suspected disease caused by N. meningitidis; History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
* Significant acute or chronic infection within the previous 7 days or axillary temperature major or equal to38 degrees within the previous day;
* Antibiotics within 6 days prior to enrollment;
* Any serious chronic or progressive disease;
* Known or suspected impairment or alteration of the immune system;
* Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation.

Ages: 2 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged 2 to 14 months selected to participate in clinical trials assessing the safety and immunogenicity of 4 component meningococcal serogroup B vaccine (4CMenB) in Austria, Belgium, Czech Republic, Finland, Germany, Italy, Spain, United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 4535 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Fever | AT RISK INTERVAL 4CMenB and inactivated routine vaccines (InRV) : Onset 24 hours following immunization (post-Imm). MMRV: Onset day 5 to day 13 post-Imm.CONTROL INTERVAL 4CMenB and InRV : Onset day 4 to 7post-Imm . MMRV: Onset day 0 to 4 post-Imm
  Temperature ≥ 38°C
Systemic reactions other than fever | AT RISK INTERVAL 4CMenB and InRV : Onset 24 hours post-Imm. MMRV: Onset day 5 to day 13 post-Imm.CONTROL INTERVAL 4CMenB and InRV : Onset day 4 to 7post-Imm . MMRV: Onset day 0 to 4 post-Imm
  systemic signs/symptoms (e.g. change in eating habits, sleepiness, unusual crying, vomiting, diarrhea, irritability…) without signs of localized infection (respiratory, urinary, etc...).
Fever or systemic reactions other than fever | AT RISK INTERVAL 4CMenB and InRV : Onset 24 hours post-Imm. MMRV: Onset day 5 to day 13 post-Imm.CONTROL INTERVAL 4CMenB and InRV : Onset day 4 to 7post-Imm . MMRV: Onset day 0 to 4 post-Imm
  all systemic signs/symptoms including fever (Temperature ≥ 38°C)
Injection site reactions | AT RISK INTERVAL all injection site reactions regardless of their delay of onset. Baseline (CONTROL) risk null.

CONTACTS AND LOCATIONS:
Overall Officials: Gaston De Serres, MD, PhD, Principal Investigator — CHU de Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gossger N, Snape MD, Yu LM, Finn A, Bona G, Esposito S, Principi N, Diez-Domingo J, Sokal E, Becker B, Kieninger D, Prymula R, Dull P, Ypma E, Toneatto D, Kimura A, Pollard AJ; European MenB Vaccine Study Group. Immunogenicity and tolerability of recombinant serogroup B meningococcal vaccine administered with or without routine infant vaccinations according to different immunization schedules: a randomized controlled trial. JAMA. 2012 Feb 8;307(6):573-82. doi: 10.1001/jama.2012.85. PMID 22318278
- [Background] Vesikari T, Esposito S, Prymula R, Ypma E, Kohl I, Toneatto D, Dull P, Kimura A; EU Meningococcal B Infant Vaccine Study group. Immunogenicity and safety of an investigational multicomponent, recombinant, meningococcal serogroup B vaccine (4CMenB) administered concomitantly with routine infant and child vaccinations: results of two randomised trials. Lancet. 2013 Mar 9;381(9869):825-35. doi: 10.1016/S0140-6736(12)61961-8. PMID 23324563
- [Background] Baker MA, Lieu TA, Li L, Hua W, Qiang Y, Kawai AT, Fireman BH, Martin DB, Nguyen MD. A vaccine study design selection framework for the postlicensure rapid immunization safety monitoring program. Am J Epidemiol. 2015 Apr 15;181(8):608-18. doi: 10.1093/aje/kwu322. Epub 2015 Mar 13. PMID 25769306
- [Derived] Zafack JG, Bureau A, Skowronski DM, De Serres G. Adverse events following immunisation with four-component meningococcal serogroup B vaccine (4CMenB): interaction with co-administration of routine infant vaccines and risk of recurrence in European randomised controlled trials. BMJ Open. 2019 May 19;9(5):e026953. doi: 10.1136/bmjopen-2018-026953. PMID 31110098